CLINICAL TRIAL: NCT05505110
Title: MOdification Of THe Early-Life Respiratory Microbiome Through Vaginal SEEDing
Acronym: MOTHER SEED
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Christian Rosas-Salazar, Assistant Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 220799; K23HL148638 (NIH)
Record Dates: First submitted 2022-08-12; First posted 2022-08-17 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: C-section; Vaginal Seeding; Respiratory; Microbiome
Keywords: C-section; Vaginal seeding; Respiratory; Microbiome

STUDY DESIGN:
Intervention Model Description: This is a single-center, parallel-arm, blind, sham-controlled, feasibility RCT to be conducted in healthy cesarean-born children.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, the principal investigator (PI), co-investigators, data manager, and the lead biostatistician will be blinded to the actual group assignment until all statistical analyses of the data required to meet the primary and co-primary endpoints have occurred. The Data and Safety Monitoring Board will remain unmasked to actual group allocation throughout the pre-specified blinding period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Active Comparator): Vaginal Seeding
  Interventions: Biological: Vaginal Seeding
- Control Group (Sham Comparator): Sterile Swab
  Interventions: Other: Sterile Swab

INTERVENTIONS:
Biological: Vaginal Seeding — Following birth by C-section and immediately after the initial newborn care by the general pediatric team, children randomized to the intervention group will have their nasal cavity swabbed with maternal vaginal secretions.
  Arms: Intervention Group
Other: Sterile Swab — Following birth by C-section and immediately after the initial newborn care by the general pediatric team, children randomized to the control group will have their nasal cavity swabbed with a sterile swab.
  Arms: Control Group

SUMMARY:
This is a single-center, parallel-arm, blind, sham-controlled, feasibility randomized controlled trial (RCT) to be conducted in healthy cesarean-born children. Eligible children will be randomized 1:1 to have their nose swabbed with either maternal vaginal secretions or a sterile swab (intervention vs. control group, respectively). The main hypothesis is that conducting an RCT assessing the utility of vaginal seeding in modifying the early-life upper respiratory tract (URT) microbiome of children born by cesarean section (C-section) is feasible and that the intervention is safe.

DETAILED DESCRIPTION:
Eligible children will be randomized 1:1 to have their nose swabbed with either maternal vaginal secretions or a sterile swab (intervention vs. control group, respectively). The procedure will be performed following birth by C-section and immediately after the initial newborn care by the general pediatric team. The mother and child will then receive usual medical care as determined by their health care providers. Follow-up will occur at multiple time points during the child's first 6 months of life. One planned interim analysis to assess the safety of the procedure will be conducted.

The intervention aims to transfer the maternal vaginal microbiome to the nasal cavity of cesarean-born children at birth (i.e., vaginal seeding of the URT). Hence, the intervention simply attempts to replicate the natural exposure to maternal vaginal secretions during vaginal delivery in children born by C-section.

ELIGIBILITY:
Inclusion Criteria:

For the mother:

* Female 18-40 years of age who is in good general health, is fully able to provide consent to participate in the study, anticipates being available for the duration of the study, and is willing to comply with all study procedures
* Singleton pregnancy
* Completed ≧3 prenatal care visits at Vanderbilt University Medical Center (any facility)
* Having rectovaginal swabs collected at ≧36 weeks of gestation to screen for Group B Streptococcus (GBS) as part of prenatal screening tests
* Having a scheduled (planned or non-emergency) C-section at Vanderbilt University Medical Center (main campus only)
* No intent to relocate outside the middle Tennessee region within 12 months of recruitment

For the child:

* Estimated gestational age ≧37 weeks
* Birth weight ≧2,500 grams

Exclusion Criteria:

For the mother:

* Past medical history of any of the following:

  * Previous child with GBS infection or prior positive GBS testing
  * Hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection
  * Genital herpes simplex virus (HSV) infection, genital herpetic lesions, or prior positive genital HSV testing
  * Genital human papilloma virus (HPV) infection, genital HPV lesions, or prior positive genital HPV testing
  * Diabetes type I or type II
* Laboratory evidence during the current pregnancy of any of the following:

  * GBS bacteriuria in urine samples collected at any time (performed as standard of care)
  * GBS colonization in rectovaginal swabs collected at ≧36 weeks of gestation (performed as standard of care)
  * Chlamydia, trichomoniasis, or gonorrhea in urine samples collected at ≧36 weeks of gestation (performed as part of the screening procedures for this study)
  * Hepatitis B, hepatitis C, HIV, or syphilis in blood samples collected at ≧36 weeks of gestation (performed as part of the screening procedures for this study)
* Uncontrolled gestational diabetes
* Any serious obstetric disease (e.g., preeclampsia with severe features, placental abruption or severe bleeding, or thromboembolic disease) as deemed by the PI or co-investigators
* Prior abnormal Pap smear
* C-section scheduled for a genitourinary infection that would have interfered with vaginal delivery (e.g., genital herpetic lesions)
* Lack of available prenatal screening tests
* Use of systemic (i.e., oral, intramuscular, or intravenous) antibiotics in the 4 weeks prior to delivery (except for those being administered as part of the C-section)
* Use of systemic (i.e., oral, intramuscular, or intravenous) immunosuppressive, biologic, or chemotherapeutic agents in the 3 months prior to delivery (except for systemic immunosuppressive agents not being used for their immunosuppressive effects [e.g., prenatal intramuscular beclomethasone for fetal lung maturation])
* Fever (≧100.4°F [38°C]) in the 72 hours prior to delivery
* Symptoms (e.g., dysuria, pruritus, or discharge) suggestive of a genitourinary infection (e.g., bacterial vaginosis, vaginal yeast infection, chorioamnionitis, or urinary tract infection) on the day of delivery
* Symptoms (e.g., pain, tenderness, tingling, burning, itching, or swollen lymph nodes) suggestive of genital HSV infection on the day of delivery
* Other symptoms (e.g., new-onset rhinorrhea, sore throat, cough, body aches, chills, nausea, vomiting, or diarrhea) suggestive of an acute infectious disease on the day of delivery
* Physical exam findings (e.g., fever [≧100.4°F (38°C)] or vesicles, warts, or ulcers in the genital, perineal, or anal region) suggestive of a genitourinary infection on the day of delivery (performed as part of the screening procedures for this study if not performed as standard of care)
* Maternal vaginal pH>4.5 on the day of delivery (performed as part of the screening procedures for this study)
* Need for a switch from a scheduled C-section to an emergency C-section
* Prelabor prolonged rupture of membranes (i.e., ≧18 hours prior to delivery)
* Pregnancy as the result of an assisted reproductive technology or surrogacy
* Participation in another clinical trial that involves an intervention that could impact the quality or interpretation of the study data as deemed by the PI or co-investigators
* Other past or current medical problems that could compromise the safety of participants, interfere with their ability to comply with study requirements, or impact the quality or interpretation of the study data as deemed by the PI or co-investigators

For the child:

* Need for neonatal measures outside routine clinical care (i.e., drying, tactile stimulation, bulb syringe or catheter suction of nose and mouth, or temperature maintenance) in the delivery room
* Transfer to the neonatal intensive care unit immediately after delivery
* Thick particulate meconium noted during delivery
* Physical exam findings (e.g., tachypnea, nasal flaring, retractions, cyanosis, or grunting) suggestive of neonatal acute respiratory distress immediately after delivery (performed as part of the screening procedures for this study)
* Prenatal diagnosis of a serious genetic, respiratory, cardiovascular, or neurological disease
* Prenatal diagnosis of intrauterine growth restriction
* Prenatal diagnosis of a major congenital anomaly (e.g., cleft lip or palate, cystic hygroma, or giant omphalocele)
* Participation in another clinical trial that involves an intervention that could impact the quality or interpretation of the study data as deemed by the PI or co-investigators
* Other past or current medical problems that could compromise the safety of participants, interfere with their ability to comply with study requirements, or impact the quality or interpretation of the study data as deemed by the PI or co-investigators

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2028-08-10 (Estimated); Study Completion 2028-08-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the RCT | Six months following randomization
  The study will be considered "definitively feasible as proposed," "possibly feasible as proposed," or "not feasible as proposed" based on eligibility, consent, enrollment, and loss to follow-up rates, which could be used as preliminary data to inform the design of a future phase II RCT. For this study, "enrolled" will be defined as consented and screened, with eligibility verified, and the eligibility, consent, enrollment, and loss to follow-up rates will be calculated using the following formulas: 1) eligibility rate = number of participants who are eligible*100 / number of participants pre-screened, 2) consent rate = number of participants who provide consent*100 / number of participants who are eligible, 3) enrollment rate = number of participants who are enrolled*100 / number of participants consented and who complete screening procedures, and 4) loss to follow-up = number of participants who did not complete the end-of-study visit*100 rate / number of participants randomized.
Safety of the intervention | Six months following randomization
  To be determined by the number of adverse events, serious adverse events, and unanticipated problems throughout the study, as defined using the standards set forth in the National Cancer Institute's - Common Terminology Criteria (NCI-CTCAE) for AEs version 4.0 and the United States Department of Health and Human Services - Reviewing and Reporting Unanticipated Problems Involving Risks to Subjects or Others and Adverse Events: Office for Human Research Protections Guidance 2007

SECONDARY OUTCOMES:
Timing of the intervention | Immediately following administration of the intervention
  The number of minutes after birth when the intervention is performed.
Proportion of in-person study visits completed | Six months following randomization
  The total number of in-person study visits completed by all participants*100 / total number of in-person visits expected for all participants for each study time point.
Common microbial ecology metrics of the maternal vaginal microbiome and of the early-life URT microbiome | At each study time point (birth, ~2 days, ~5 days, ~4 weeks, and ~6 months of age) and over time (longitudinally from birth to age 6 months)
  The comparisons of the maternal vaginal microbiome on the day of delivery between study groups will be conducted using alpha-diversity (e.g., observed taxa, Shannon index, and Simpson indices), beta-diversity (e.g., Bray-Curtis, Jaccard, weighted UniFrac, and unweighted UniFrac indices), and differential abundance (at the amplicon sequence variant, genus, and/or family level) analyses. The early-life URT microbiome at each time point and over time will be compared between study groups using similar microbial ecology metrics. In pre-specified analyses, we will also compare the presence and abundance of the genus Lactobacillus and the predominant Lactobacillus amplicon sequence variants in the URT of children at each time point and over time between study groups, as this is the predominant taxa of the maternal vaginal microbiome during pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Rosas-Salazar, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified next-generation sequencing data generated as part of this study will be deposited into NIH-sponsored or other scientific repositories immediately following a publication. Other de-identified individual participant data (IPD) that underlie the results reported in a manuscript will be shared with other parties upon request beginning 12 months and ending 36 months following a publication. In addition, the study protocol and informed consent documents will be uploaded to clinicaltrials.gov no later than 60 days after the end-of-study visit of the last enrolled participant.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified next-generation sequencing data generated as part of this study will be deposited into NIH-sponsored or other scientific repositories immediately following a publication. Other de-identified IPD that underlie the results reported in a manuscript will be shared with other parties upon request beginning 12 months and ending 36 months following a publication. In addition, the study protocol and informed consent documents will be uploaded to clinicaltrials.gov no later than 60 days after the end-of-study visit of the last enrolled participant.
Access Criteria: Individual requests for de-identified IPD sharing from other parties will be evaluated and approved by the PI. For this, the requesting party will need to provide a methodologically sound proposal, obtain approval from their Institutional Review Board, and sing a data sharing agreement. De-identified IPD will be mainly shared for the purpose of conducting a systematic review with meta-analysis, but other studies will be evaluated on a case-by-case basis.